CLINICAL TRIAL: NCT00212017
Title: The Japan Working Group for the Assessment That the Alpha-glucosidase Inhibitor Blocks Cardiac Events in Patients With Myocardial Infarction and IGT
Brief Title: Assessment of an Alpha-glucosidase Inhibitor to Block Cardiac Events in Patients With MI and IGT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We obtained the final results due to the interim analysis.
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Collaborators: Ministry of Health, Labor and Welfare (Japan) (Unknown)
Responsible Party: Principal Investigator, Masafumi Kitakaze, Director, National Cerebral and Cardiovascular Center, Japan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CSSCJ-3; UMIN_ID:C000000090
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Impaired Glucose Tolerance; Myocardial Infarction
Keywords: IGT; Myocardial Infarction; alpha-glucosidase inhibitor; re-infarction prevention
MeSH Terms: conditions — Glucose Intolerance; Myocardial Infarction | interventions — voglibose; Diet; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, open, blinded-endpoint study
Who Masked: Outcomes Assessor
Masking Description: This is an open and blinded-endpoint study

ARMS (2):
- the voglibose group (Active Comparator): Participants in the voglibose group were administered a voglibose tablet (0.2 mg) three times daily before meals.
  Interventions: Drug: voglibose
- the control group (Active Comparator): Participants assigned to the control group were treated only with diet and exercise therapy.
  Interventions: Behavioral: diet and exercise therapy

INTERVENTIONS:
Drug: voglibose
  Arms: the voglibose group
Behavioral: diet and exercise therapy
  Arms: the control group

SUMMARY:
The purpose of this study is to evaluate whether an alpha-glucosidase inhibitor, a drug for the suppression of postprandial hyperglycemia, could reduce the recurrence of myocardial infarction in patients with impaired glucose tolerance (IGT) and old myocardial infarction.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is a well-established risk factor for coronary heart disease and atherosclerotic change in the coronary artery develops subclinically in a state of impaired glucose tolerance (IGT). Recently postprandial hyperglycemia as a feature of impaired glucose tolerance is recognized as a significant risk factor for coronary heart disease. So we designed a prospective randomized multi-center trial named Assessment of an α-glucosidase-inhibitor to Block Cardiac Events in Patients With Myocardial Infarction and IGT (ABC study) to evaluate whether an α-Glucosidase Inhibitor, a drug for the suppression of postprandial hyperglycemia, could reduce the recurrence of myocardial infarction in patients with IGT and old myocardial infarction.

100 hospitals will participate in the ABC study. Patients with IGT who have a history of prior myocardial infarction are randomly allocated to receive α-Glucosidase Inhibitor (voglibose) or a standard diet and exercise treatment. The number of patients to be recruited is 3000 and this study will continue for at least 2 years. The primary end-points are:

1. cardiovascular mortality and
2. hospitalization for cardiovascular events.

Effects in suppression of new diabetes development will also be evaluated.

We should recognize IGT as an important therapeutic target to decrease the recurrence of cardiovascular events. The ABC study, a large scale multi-center trial in Japan, will provide us with new evidence on how to treat IGT patients with prior myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

1. Impaired glucose tolerance
2. History of myocardial infarction

Exclusion Criteria:

1. Type I diabetes
2. History of coronary artery bypass graft
3. Severe liver and/or kidney dysfunction
4. History of allergic response to drugs
5. Arteriosclerosis obliterans

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
the time till the first cardiovascular composite endpoint of death from cardiovascular death, and hospitalization due to nonfatal myocardial infarction, nonfatal unstable angina[16], nonfatal stroke, or treatment with coronary revascularisation | May 2005 and June 2012
  the time till the first cardiovascular composite endpoint of death from the time till the first cardiovascular composite endpoint of death from cardiovascular death, and hospitalization due to nonfatal myocardial infarction, nonfatal unstable angina[16], nonfatal stroke, or treatment with coronary revascularisation

SECONDARY OUTCOMES:
All cause mortality | May 2005 and June 2012
  All cause death
Hospitalization due to coronary artery disease | May 2005 and June 2012
  Hospitalization due to coronary artery disease
Progression of IGT to diabetes | May 2005 and June 2012
  Progression of IGT to diabetes
Development or deterioration of either hypertension or hyperlipidemia | May 2005 and June 2012
  Development or deterioration of either hypertension or hyperlipidemia
Deterioration of renal function | May 2005 and June 2012
  Deterioration of renal function
Hospitalization due to cerebrovascular disease | May 2005 and June 2012
  Hospitalization due to cerebrovascular disease
Hospitalization due to heart failure | May 2005 and June 2012
  Hospitalization due to heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Masafumi Kitakaze, MD, PhD, Study Chair — National Cerebral and Cardiovascular Center, Japan
Locations (1):
- National Cardiovascular Center, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Asakura M, Kim J, Asanuma H, Hamasaki T, Tsukahara K, Higashino Y, Ishikawa T, Nakama Y, Koba S, Maruyama Y, Tsujimoto M, Himeno H, Ohkusa T, Fujino S, Shimizu M, Endo T, Yoda S, Muroya T, Murohara T, Ohte N, Suzuki H, Kohno T, Fukui K, Shiono T, Takase H, Uzui H, Nagai Y, Hashimoto Y, Ikeda S, Mizuno S, Tamita K, Fujita M, Satake K, Kinoshita Y, Nunohiro T, Sakagami S, Higaki J, Morii I, Sawada R, Hiasa Y, Shigemasa T, Nakahama M, Sata M, Doi O, Ueda T, Yamada T, Yamanouchi T, Yamaguchi H, Morita Y, Hayashi H, Kitakaze M; ABC investigators. Does Treatment of Impaired Glucose Tolerance Improve Cardiovascular Outcomes in Patients with Previous Myocardial Infarction? Cardiovasc Drugs Ther. 2017 Aug;31(4):401-411. doi: 10.1007/s10557-017-6740-3. PMID 28779371